CLINICAL TRIAL: NCT07114562
Title: A Prospective, Interventional, Evaluator-Blinded, Multi-Center Study for the Assessment of the Safety and Performance of Epicare for the Treatment of Periorbital Wrinkles
Brief Title: Evaluation of the Safety and Performance of Epicare for the Treatment of Periorbital Wrinkles
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laser team Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PL-001
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Periorbital Wrinkles
Keywords: Wrinkles; Periorbital wrinkles; Aesthetic dermatology; Laser resurfacing; Fractional thulium laser; Epicare

STUDY DESIGN:
Intervention Model Description: Allocation: Non-Randomized
  Intervention Model: Single Group Assignment (all participants receive Epicare treatment)
  Masking: Evaluator-Blinded (photographs assessed by blinded independent reviewers)
  Primary Purpose: Treatment
Masking Description: Evaluator-Blinded (photograph reviewers; subjects and investigators unblinded)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epicare treatment arm (Experimental): All participants will receive treatment with the Epicare fractional nano-thulium (Tm:YAP, 1938 nm) laser device for the reduction of periorbital wrinkles.
  Interventions: Device: Epicare

INTERVENTIONS:
Device: Epicare — All participants will receive treatment with the Epicare fractional nano-thulium (Tm:YAP, 1938 nm) laser device for the reduction of periorbital wrinkles.

SUMMARY:
This is a prospective, interventional, evaluator-blinded, multi-center clinical study designed to assess the safety and performance of the Epicare fractional nano-thulium (Tm:YAP 1938 nm) laser system for the treatment of moderate to severe periorbital wrinkles in adults aged 25-65. Up to 50 participants will receive one Epicare treatment at baseline, with an optional second treatment at Month 2 based on clinical assessment. The primary endpoint is the proportion of participants achieving at least a 1-grade improvement on the Fitzpatrick Wrinkle Classification Scale (FWCS) three months after the last treatment, as evaluated by at least 2 of 3 independent, blinded reviewers of standardized photographs.

DETAILED DESCRIPTION:
The Epicare device utilizes fractional nano-thulium (Tm:YAP 1938 nm) laser technology to create precise ablative micro-columns surrounded by adjustable coagulative zones, stimulating collagen regeneration and dermal remodeling while minimizing thermal injury and downtime. This clinical investigation will enroll 50 adults with Fitzpatrick skin types I-V and bilateral, approximately symmetrical periorbital wrinkles (FWCS 4-9).

Participants undergo standardized photography, FWCS scoring, GAIS evaluations, pain assessment (VAS), downtime assessments, and adverse event monitoring. Treatment #1 occurs at baseline and an optional Treatment #2 may be performed at Month 2. The End-of-Study visit occurs 3 months after the last treatment (Month 5 for two-treatment participants).

The study evaluates performance outcomes (FWCS, GAIS, satisfaction) and safety (device-related adverse events). No interim analysis is planned. Data will be analyzed descriptively. This pivotal clinical investigation is intended to establish the safety and performance of the Epicare device for aesthetic treatment of periorbital wrinkles.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 25-65 years of age, in general good health.
* Seeking a reduction in the appearance of periorbital wrinkles.
* Bilateral and approximately symmetrical periorbital wrinkles with a Fitzpatrick Wrinkle Classification Scale (FWCS) score 4-9, as assessed by the treating investigator.
* Fitzpatrick skin type I-V.
* Able to understand the study requirements and sign an EC/IRB-approved informed consent form prior to any study procedures.
* Willing and able to comply with the treatment and follow-up schedule, pre- and post-treatment instructions, and allow standardized photography.
* Willing to withhold additional aesthetic therapies to the treatment area (e.g., fillers, resurfacing procedures) for the entire study duration.

Exclusion Criteria:

* Known bleeding disorder (e.g., thrombocytopenia, thrombasthenia, von Willebrand's disease).
* Immunocompromised or immunosuppressed (e.g., AIDS, HIV, or immunosuppressive therapy).
* Planned or recent use of anti-platelets, anti-coagulants, thrombolytics, ACE inhibitors, vitamin E, or anti-inflammatory drugs from 1 week prior to 1 month after treatment.
* Systemic corticosteroid or anabolic steroid use within 30 days prior to enrollment (standard inhaled/nasal corticosteroids are permitted).
* Use of weight loss medications before or during the study.
* History of chronic or recurrent infection or inflammation that would preclude participation.
* Severe allergies with history of anaphylaxis.
* History of malignancy within 5 years prior to enrollment.
* Infection, inflammation, or active dermatologic disease in the face.
* Pregnant, breastfeeding, or planning pregnancy during the study; women of childbearing potential not using reliable contraception for ≥3 months prior and throughout the study.
* Exposure to an investigational drug or device within 3 months prior to enrollment or during the study.
* Prior permanent facial injections (e.g., silicone, grafting) or any upper-face surgery.
* Neurotoxin treatments in the upper face within 6 months prior to enrollment.
* Semi-permanent filler (e.g., collagen, CaHA) or any dermal filler (e.g., hyaluronic acid) in the upper face within 18 months prior to enrollment.
* Any active or passive implant in the treatment area (metallic, silicone, electronic, or injected chemical substance).
* Initiation of over-the-counter anti-wrinkle products (e.g., alpha-hydroxy acids) or prescription treatments (e.g., Retin-A, micro-dermabrasion, chemical peels) within 4 weeks prior to enrollment or planned use during the study.
* Occupations involving continuous or routine sun exposure (e.g., lifeguards, outdoor workers).
* History of smoking within the past 5 years.
* Planned bariatric surgery or recent drastic weight loss.
* Unstable body weight during the study.
* Any other medical condition, laboratory abnormality, or investigator judgment that could affect compliance, safety, or data integrity.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Fitzpatrick Wrinkle Classification Scale (FWCS) improvement after three months from last treatment. | 3 months post-Treatment #2
  Proportion of participants achieving ≥1-grade improvement on the Fitzpatrick Wrinkle Classification Scale (FWCS) three months after Treatment #2, evaluated by ≥2 of 3 independent blinded reviewers.

SECONDARY OUTCOMES:
Physician-Reported GAIS Improvement | 3 months post-Treatment #2
  Physician Global Aesthetic Improvement Scale (P-GAIS): 5-point ordinal scale (1 = Worse, 2 = No Change, 3 = Improved, 4 = Much Improved, 5 = Very Much Improved).
Physician-Reported FWCS Improvement | 3 months post-Treatment #2
  Fitzpatrick Wrinkle Classification Scale (FWCS): 0-9 grading scale assessing the severity of periorbital wrinkles.Change from baseline in FWCS, assessed by the investigator.
Subject-Reported GAIS | 3 months post-Treatment #2
  Subject Global Aesthetic Improvement Scale (S-GAIS): 5-point ordinal scale reported by the participant, reflecting perceived aesthetic improvement (1 = Worse, 2 = No Change, 3 = Improved, 4 = Much Improved, 5 = Very Much Improved).
Subject-Reported S-GSQ | 3 months post-Treatment #2
  Subject Global Satisfaction Questionnaire (S-GSQ): Structured questionnaire assessing the participant's overall satisfaction with treatment results and willingness to recommend/undergo treatment again
Pain Assessment Using Visual Analog Scale (VAS) After Each Treatment | Immediately post-procedure at each treatment visit
  Visual Analog Scale (VAS) for pain: 0-10 scale (0 = no pain, 10 = worst imaginable pain).Participants rate the maximum procedural pain immediately after treatment.
  Recorded in the CRF for safety and tolerability evaluation.
Subjective Downtime Assessment After Each Treatment | Collected at Week 1 post-treatment follow-up visits for each treatment session.
  Subject Downtime Questionnaire evaluating perceived post-treatment recovery and any restrictions to daily activities, typically rated on a categorical scale (e.g., None, Mild, Moderate, Severe).

CONTACTS AND LOCATIONS:
Overall Officials: Yoav Gronovich, Dr., Principal Investigator — Shaare Zedek Medical Center; Avshalom Shalom, Prof., Principal Investigator — Meir Medical Center

IPD SHARING:
Plan to Share IPD: No